CLINICAL TRIAL: NCT02082496
Title: Exploration of the Physiological Effect of GLP-1 in Obese Adults Diagnosed With Obesity Causing Genetic Mutations
Brief Title: GLP-1 Response and Effect in Individuals With Obesity Causing Genetic Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Eva Pers Winning Iepsen, M.D., University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MC4R-2014
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Obesity
Keywords: Obesity; Obesity Genetics; GLP-1; GLP-1 Receptor Agonists
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Experimental): 4 months intervention with Liraglutide 3.0 mg daily as subcutanous injection
  Interventions: Drug: Liraglutide
- Case Group (Experimental): 4 months intervention with Liraglutide 3.0 mg daily as subcutanous injection
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — S.c. liraglutide 3.0mg once daily
  Other Names: Victoza, Novo Nordisk A/S in DK-2880 Bagsvaerd; Serial number:76477425; International code name: 005; US Class Codes: 006, 018, 044, 046, 051, 052

SUMMARY:
The obesity epidemic is attributable to dietary and behavioral trends acting on a person's genetic makeup to determine body mass and susceptibility to obesity-related diseases. Furthermore, common forms of obesity have a strong hereditary component and many genetic pathways that contribute to obesity have already ben identified.

Glucagon-like peptide-1 (GLP-1) is an incretin hormone that potentiates glucose-stimulated insulin secretion. However, GLP-1 also acts as an appetite-inhibiting hormone affecting the appetite center in the hypothalamus. Today, GLP-1 receptor agonists are available for the treatment of type 2 diabetes, and their treatment potential in obesity is an area of active research.

The aim of this study is to explore if the appetite inhibiting effect of GLP-1 is intact in people diagnosed with obesity causing genetic disorders and to investigate the physiological role of GLP-1 on food intake and appetite regulation in this group.

DETAILED DESCRIPTION:
* Exploration of the physiological role of GLP-1 concerning food intake and appetite regulation in obese adults diagnosed with obesity related genetic disorders.
* Assessment of the effect of GLP-1 on body composition, bone mineral density, energy expenditure, cardiac function, glucose tolerance, insulin sensitivity, lipid concentrations and neuroendocrine function.
* Assessment of the impact of the leptin induced adaptive thermogenesis response in the weight reduced study participants.
* Investigating the alteration of the composition of gut bacteria as well as subjective ratings of satiety and hunger before after supplement with GLP-1.

ELIGIBILITY:
Inclusion Criteria:

* BMI above 28 (kg/m2)
* age 18-65 years
* otherwise healthy

Exclusion Criteria:

* pregnancy or breastfeeding
* Type 2 Diabetes
* suffering from severe medical conditions

Recruitment for this study finished November 2015

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Difference in insulin levels in reponse to GLP-1 RA treatment in obese genetic mutation carriers vs obese controls | 4 months intervention
  pmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Jens J Holst, Professor, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Biomedical Sciences, Copenhagen, Denmark